CLINICAL TRIAL: NCT03759340
Title: Open-Label Study of ATI-502 Topical Solution for the Treatment of Alopecia Areata (AA), Alopecia Universalis (AU) and Alopecia Totalis (AT)
Brief Title: ATI-502 Topical Solution for the Treatment of Alopecia Areata (AA), Alopecia Universalis (AU) and Alopecia Totalis (AT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-502-AA-203
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Results first posted 2020-09-17 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Alopecia Areata; Alopecia Universalis; Alopecia Totalis
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: This Phase 2, multicenter, open-label study will evaluate the safety, tolerability, efficacy, and durability of efficacy of ATI-502 Topical Solution, 0.46% for the treatment of alopecia areata (AA), alopecia universalis (AU) and alopecia totalis (AT) in adult subjects who completed 24 weeks of treatment with ATI-501 Oral Suspension or Placebo Suspension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATI 502 0.46% Topical Solution (Experimental): Subjects will apply ATI-502 Topical Solution, 0.46% twice-daily for 24 weeks followed by a 4-week post-treatment follow up period.
  Interventions: Drug: ATI 502 0.46% Topical Solution

INTERVENTIONS:
Drug: ATI 502 0.46% Topical Solution — apply ATI-502 Topical Solution, 0.46% Twice a day (BID) to the entire scalp and if applicable, the eyebrow(s)

SUMMARY:
This is an open label study of ATI-502 Topical Solution for the treatment of AA, AU, and AT with the following goals:

* To assess the safety, tolerability, and efficacy of ATI-502 Topical Solution in subjects with AA, AU or AT following 24 weeks of treatment with ATI-501 Oral Suspension or Placebo Suspension.
* To assess the ability of ATI-502 Topical Solution to maintain or improve hair regrowth in subjects previously treated with ATI-501 Oral Suspension or Placebo Suspension.

DETAILED DESCRIPTION:
This Phase 2, multicenter, open-label study will evaluate the safety, tolerability, efficacy, and durability of efficacy of ATI-502 Topical Solution, 0.46% for the treatment of alopecia areata (AA), alopecia universalis (AU) and alopecia totalis (AT) in adult subjects who completed 24 weeks of treatment with ATI-501 Oral Suspension or Placebo Suspension.

Subjects who complete 24 weeks of active treatment with ATI-501 Oral Suspension or Placebo Suspension in study ATI-501-AUAT-201 will be assessed for eligibility to enter the study. At Visit 9 in study ATI-501-AUAT-201, subjects who did not experience any adverse events (AEs), serious adverse events (SAEs), or tolerability issues that met study discontinuation criteria in study ATI-501-AUAT-201 and who in the opinion of the investigator are capable of re-growing or maintaining scalp hair and meet the entry criteria are eligible to enroll in this open-label study.

Enrolled subjects will apply ATI-502 Topical Solution, 0.46% BID to the entire scalp and if applicable, the eyebrow(s) and return for safety and efficacy assessments as detailed in the Schedule of Assessments (Table 3). Assessment of response to treatment will be performed at Week 4, Week 8, Week 16, Week 24, and post-treatment Week 28. Safety and tolerability will be evaluated at each study visit by assessment of adverse events, clinical laboratory tests, and vital signs, and at Week 24, and physical examination findings

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to be eligible for participation in the study:

  1. Subject must be able to comprehend and willing to sign the Informed Consent Form (ICF).
  2. Male or non-pregnant, non-nursing female ≥ 18 years old at the time of informed consent.
  3. Subject has completed 24 weeks of treatment and the assessments for Visit 9 in study ATI-501-AUAT-201.
  4. Subject has not experienced any AEs, SAEs or tolerability issues that met study discontinuation criteria in ATI-501-AUAT-201.
  5. Subject is capable of regrowing scalp hair or maintaining prior scalp hair regrowth from ATI-501-AUAT-201 in the opinion of the investigator.
  6. If a woman of childbearing potential (WOCBP), must have a negative urine pregnancy test at Visit 1 and agree to: use a highly effective method of birth control for the duration of the study; not be planning a pregnancy during the study duration and use contraception for 30 days after last application of study medication. (Refer to Section 8.4).
  7. Be in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of the subject or which might expose the subject to an unacceptable risk by study participation.
  8. Be willing to maintain the same general hair style throughout the study period. Subjects who shave their scalp must be willing to refrain from shaving their scalp for at least one week or longer prior to each study visit, as determined by the investigator based on visible scalp hair growth. Hair trimming outside the treatment areas to maintain the current hair style is permitted.
  9. Be willing and able to follow all study instructions and to attend all study visits.
  10. Sexually active male subjects must agree to use a barrier method of contraception from the first application of study medication to at least 30 days after the last application of study medication.

Exclusion Criteria:

* Subjects are excluded from this study if any 1 or more of the following criteria is met:

  1. Any study medication discontinuation criteria are met during participation in study ATI-501-AUAT-201.
  2. Females who are nursing, pregnant, or planning to become pregnant for the duration of the study and up to 30 days after the last application of study medication.
  3. The presence of a permanent or difficult to remove hairpiece or wig that will, in the opinion of the investigator, interfere with study assessments if not removed at each visit.
  4. Sensitivity to any of the ingredients in the study medications.
  5. Unwillingness to refrain from weaves, hair extensions, or shaving of the scalp for at least one week or longer prior to each study visit, as determined by the investigator based on visible scalp hair growth the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Aclaris Investigator Site, Rogers, Arkansas
  - Aclaris Investigator Site, Denver, Colorado
  - Aclaris Investigator Site, Boynton Beach, Florida
  - Aclaris Investigator Site, Snellville, Georgia
  - Aclaris Investigator Site, Clinton Township, Michigan
  - Aclaris Investigator SIte, Detroit, Michigan
  - Aclaris Investigator Site, Fridley, Minnesota
  - Aclaris Investigator Site, Minneapolis, Minnesota
  - Aclaris Investigator Site, Saint Joseph, Missouri
  - Aclaris Investigator Site, Omaha, Nebraska
  - Aclaris Investigator Site, Las Vegas, Nevada
  - Aclaris Investigator Site, New York, New York
  - Aclaris Investigator Site, Rochester, New York
  - Aclaris Investigator Site, Portland, Oregon
  - Aclaris Investigator Site, Greenville, South Carolina
  - Aclaris Investigator Site, Knoxville, Tennessee
  - Aclaris Investigational Site, Nashville, Tennessee
  - Aclaris Investigational Site, Austin, Texas
  - Aclaris Investigator Site, Houston, Texas
  - Aclaris Investigator Site, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- ATI-502 0.46% Topical Solution: Subjects will apply ATI-502 Topical Solution, 0.46% twice-daily for 24 weeks followed by a 4-week post-treatment follow up period.
  ATI-502 0.46% Topical Solution: apply ATI-502 Topical Solution, 0.46% Twice a day (BID) to the entire scalp and if applicable, the eyebrow(s).
Period: Overall Study
Arm/Group | ATI-502 0.46% Topical Solution
Started | 56
Completed | 0
Not Completed | 56
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 15
Not completed — Study Terminated by Sponsor | 38

BASELINE CHARACTERISTICS:
Population: ATI-50002 0.46% Topical Solution applied twice daily.
Arm/Group | ATI 502 0.46% Topical Solution
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 42
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 56
Duration of Current Alopecia Episode (years) [Mean (Standard Deviation); unit: years] | 4.5 (3.19)
Duration of Alopecia (years) [Mean (Standard Deviation); unit: years] | 12.6 (12.09)
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 2
  II - Burns Easily | 19
  III - Burns Moderately | 20
  IV - Burns Minimally | 6
  V - Rarely Burns | 8
  VI - Never Burns | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in the Severity of Alopecia Tool (SALT) Score
Description: The Severity of Alopecia Tool (SALT) score is a physician administered scale measuring the amount of scalp without any terminal hair assessed by the investigator. Possible scores range from 0 (no scalp hair loss) to 100 (complete scalp hair loss). A negative change in the SALT score over time represents hair regrowth by adding the percentage hair loss in the various areas (i.e. top, back, each side) of the scalp. For the primary endpoint, the primary efficacy variable was the mean relative percent change from the original baseline visit in study ATI-501-AUAT-201 and the SALT score at Week 24 on study ATI-502-AA-203. This represents the percentage of hair regrowth. It was calculated as the mean of the changes from baseline SALT score to the SALT score at Week 24, divided by baseline SALT score and expressed as a percentage.
Time Frame: Baseline to Week 24
Population: Only 8 of the 56 enrolled participants had efficacy measures on Day 169 (primary endpoint) of the ATI-502-AA-203 study. Based on this limited data set, the maintenance of, or new hair regrowth cannot be adequately assessed from this study.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | ATI 502 0.46% Topical Solution
Number analyzed (Participants) | 8
Percent Change from Baseline | -15.72 (35.383)

2. Secondary Outcome: Mean Relative Percent Change From Baseline SALT Score
Description: Mean Relative Percent Change from Baseline (from the current study ATI-502-AA-203) in Severity of Alopecia Tool (SALT). SALT score is on a percent scale where 0% is no hair loss and 100 % is total hair loss. A lower SALT score is a better outcome. A higher relative percent change is better.
Time Frame: Baseline to Week 24
Population: Due to the premature termination of the study, the secondary efficacy endpoint analyses were not performed.
Arm/Group | ATI 502 0.46% Topical Solution
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Subjects Achieving a SALT50 (Defined as a ≥ 50% Improvement From Baseline in SALT) by Visit
Description: Proportion of subjects achieving a SALT 50 (defined as a ≥ 50% improvement from baseline in SALT) by visit 6. SALT score is on a percent scale where 0% is no hair loss and 100 % is total hair loss.
Time Frame: Baseline to Week 24
Population: Due to the premature termination of the study, the secondary efficacy endpoint analyses were not performed.
Arm/Group | ATI 502 0.46% Topical Solution
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Subjects Achieving a SALT 75 (Defined as a ≥ 75% Improvement From Baseline in SALT) by Visit
Description: Proportion of subjects achieving SALT 75 (defined as a ≥ 75% improvement from baseline in SALT) by visit 6 SALT score is on a percent scale where 0% is no hair loss and 100 % is total hair loss. A bigger percent change is a more positive score.
Time Frame: Baseline to Week 24
Population: Due to the premature termination of the study, the secondary efficacy endpoint analyses were not performed.
Arm/Group | ATI 502 0.46% Topical Solution
Number analyzed (Participants) | 0

5. Secondary Outcome: Durability of Response
Description: Durability of response: Proportion of subjects achieving a SALT 50 or SALT 75 at Week 24 (in study ATI-501-AUAT-201) and maintaining that response at week 24 in ATI-502-AA-203 study.
Time Frame: Baseline to Week 24
Population: Due to the premature termination of the study, the secondary efficacy endpoint analyses were not performed.
Arm/Group | ATI 502 0.46% Topical Solution
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in the Physician Global Impression of Severity (PhGIS)
Description: Change from Baseline in the PhGIS by visit. The PhGIS is a 5 point scale from Mild to Extremely Severe. Mild is a better outcome.
Time Frame: Baseline to Week 24
Population: Due to the premature termination of the study, the secondary efficacy endpoint analyses were not performed.
Arm/Group | ATI 502 0.46% Topical Solution
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment Period = 24 weeks; Reporting of non-serious AEs started with each subject's first study medication application and continued until the end of the subject's last study visit. Reporting for SAEs started when the subject signed the informed consent document and continued until the end of the subject's last visit.
Arm/Group | ATI 502 0.46% Topical Solution
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 18/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI 502 0.46% Topical Solution (N=56)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Application site dryness (General disorders) | 2 (2)
Application site pruritus (General disorders) | 2 (2)
Application site rash (General disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pyuria (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2)
White blood cell count increased (Investigations) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The ATI-502-AA-203 study was terminated early due to lack of efficacy in a similarly designed study with ATI-502 Topical Solution. Due to the premature termination, the secondary efficacy analyses outlined in the protocol were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT03759340/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT03759340/ICF_001.pdf